CLINICAL TRIAL: NCT04735562
Title: Association of Plasma Thrombospondin-4 Levels and Peripheral Arterial Disease in Hemodialysis Patients
Brief Title: Thrombospondin-4 Levels and Peripheral Arterial Disease in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 109056
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Thrombospondin-4; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Peripheral arterial disease (PAD) a condition characterized by atherosclerotic occlusive disease of the lower extremities is commonly observed in patients with chronic kidney disease (CKD) patients, particularly those on dialysis. The investigators conducted detailed biomarkers such as thrombospondin and related inflammatory biomarkers for the risk of developing and presence of PAD. Thrombospondin-4 (TSP-4) is an extracellular matrix protein of the vessel wall. Despite bench evidence, its significance in the clinical setting of chronic kidney disease (CKD) is missing

Methods:

This is a cross-sectional, single-center study. A cohort of 450 patients aged 20 or over, who have been on HD for at least 3 months prior to enrollment (Dec 1, 2021) will be included. TSP-4 and TSP-1 will be measured in HD patients using a commercially available ELISA. PAD is diagnosed by the ankle-brachial index (ABI) We will measure related blood biomarkers such as serum hs-cTnT, N-terminal probrain natriuretic peptide, s-Klotho and FABP-4.

DETAILED DESCRIPTION:
Study Population and Data Source This is a cross-sectional, single-center study which will be conducted in the Dialysis Center of Tungs' Taichung MetroHarbor Hospital (TTMHH) in the coastal region of central Taiwan. A cohort of 450 patients aged 20 or over, who have been on HD for at least 3 months prior to enrollment (Dec 1, 2021) will be included. The medical charts of these patients are reviewed for eligibility identification, and should be compatible with the inclusion/exclusion criteria and enrolled in our analysis.

In this study, the diagnostic criterion for asymptomatic PAD is an ABI value lower than or equal to 0.9 with no clinical symptoms in the lower limb such as muscle discomfort or intermittent claudication. PAD is considered symptomatic if patients have an ABI ≤0.9 and clinical symptoms or if they undergo previous surgical revascularization procedures or limb amputation. The characteristics of patients will be exclude from our study were (1) baseline ABI values > 1.3 , (2) symptomatic PAD , (3) decompensated cirrhosis , (4) neoplastic diseases , (5) incomplete data, (6) receiving hemodialysis < 3 months and active infection. The baseline data such as demographics, comorbidities, anthropometrics, and relevant laboratory data, clinical diagnosis of PAD based on measurements of ABI, and medication history will be collected.

Ankle Brachial Index Measurements The ABI was measured by trained technicians using the Fukuda Vascular Screening System (VaSera VS-1000™, Fukuda Denshi Co., Ltd., Tokyo, Japan), which measures blood pressure from bilateral arm and ankle (brachial and posterior tibial arteries, resp.) simultaneously by an oscillometric method. The systolic pressure of the arm without dialysis access and the lower value of the ankle systolic pressure were used for the calculation. ABI was calculated by the ratio of the ankle systolic pressure divided by the arm systolic pressure. Of the two ABI values, respectively, calculated from the left- and right-limb measurements, the lowest value is used in this study. All participants were annually measured in a supine position after resting for at least 15 minutes and before dialysis.

In this study, ABI less than 0.90 was considered as evidence of PAD . Absence of PAD was defined as ABI between 0.90 and 1.30 . Individuals with ABI greater than 1.30 were excluded, because this indicates poorly compressible leg arteries and inability to gauge arterial perfusion accurately .

Laboratory Mesaurements Blood was drawn with EDTA anticoagulant in the morning after an overnight fast of at least 12 h before a dialysis session. The samples were separated via centrifugation (4000 rpm, 10 min) and immediately stored at -80°C for subsequent assays. Glucose, high-density lipoprotein cholesterol HDL), triglycerides and total cholesterol are all measured by standard assays using the analyzer. Low-density lipoprotein cholesterol (LDL) is measured by standard assay. Beta 2 microglobulin, high-sensitivity C-reactive protein (hsCRP) and are measuredusing standard nephelometry. Serum hs-cTnT was measured using a sandwich immunoassay method, a novel highly sensitive assay with a lower measurable limit of 3 ng/L. N-terminal probrain natriuretic peptide(NT-proBNP) is measured using a sandwich immunoassay method, the lower limits of quantification were 5 pg/mL. The serum levels of a-Klotho were measured using an enzyme linked immunosorbent assay (ELISA) system, and this assay detects circulating a-Klotho using 2 monoclonal antibodies that specifically recognize the extracellular domain of Klotho, the lower limits of quantification were 6.15 pg/mL and the intra-assay and interassay coefficients of variation of <10%. Plasma blood concentrations of FABP4 were measured by means of (sandwich) ELISA (enzyme-linked immunosorbent assay). Plasma TSP-1 and TSP-4 levels were assessed via ELISA. Calculated intra-assay and interassay coefficient of variation for TSP-4 were 9.3% and 7.7%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* A cohort of aged 20 or over, who have been on HD for at least 3 months prior to enrollment (Dec 1, 2021) will be included.

Exclusion Criteria:

* (1) baseline ABI values > 1.3 , (2) symptomatic PAD , (3) decompensated cirrhosis , (4) neoplastic diseases , (5) incomplete data, (6) receiving hemodialysis < 3 months and active infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of biomarkers of thrombospondin-4 levels | 1 years
  Plasma level of thrombospondin-4 is a biomarkers for the risk of developing and presence of PAD

SECONDARY OUTCOMES:
Ankle Brachial Index Measurements | 1 years
  Diagnostic criterion for asymptomatic PAD
Analysis of biomarkers of hs-cTnT | 1 years
  The hs-cTnT was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of N-terminal probrain natriuretic peptide | 1 years
  The N-terminal probrain natriuretic peptide was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of a-Klotho | 1 years
  The a-Klotho was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of FABP-4 | 1 years
  The FABP-4 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan